CLINICAL TRIAL: NCT04548037
Title: Assessment of Emotional Memory During Transient Global Amnesia
Acronym: EMOTICTUS
Status: Terminated | Type: Observational
Why Stopped: Departure of the principal investigator
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2019-01/CH-01
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Amnesia, Transient Global
MeSH Terms: conditions — Amnesia, Transient Global

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with transient global amnesia
  Interventions: Other: PET-CT examination
- Healthy volunteers

INTERVENTIONS:
Other: PET-CT examination — The subject is placed in supine position, the head immobilized in a headrest. The imaging sequence begins with a scout view (viewing angle 90 °, 120 kV, 20 mA), then an X-ray scan is performed for the attenuation correction (120 kV, 5 mAs per slice, pitch 0.531, collimation 40 mm , FOV 70) and diagnostic CT scan (120 kV, 100-250 mA: auto mA, pitch 0.531, 40 MM, DFOV 25, ASIR 60%, thickness 1.25 mm). Finally, the positron emission tomography is acquired: static in 3D mode for 15 minutes, 30 minutes after the injection of 18 FDG, the axial field of view is 25, the matrix in 256 x 256, OSEM reconstruction 6 iterations 24 subsets, attenuation correction, diffused, and PSF. Gaussian filter, cutoff frequency of 4. Obtaining forty-seven contiguous sections of 3.26 mm thick.
  Groups: Patients with transient global amnesia

SUMMARY:
There are few studies on the role played by emotions in transient global amnesia (TGA), in particular with regard to their impact on the functioning of memory. The study investigators wish to better understand the link between episodic memory, emotional state and psychogenic factors during TGA. It would be interesting to see if the patients suffering from TGA triggered by a psychological shock process emotional information differently from those whose TGA was triggered by an "organic" shock (physical effort, trauma, etc.). Finally, amnesic stroke is a good model for better understanding the function of the hippocampus, in particular of the CA1 region, in episodic memory.

ELIGIBILITY:
Inclusion Criteria:

* Subject with no history of transient global amnesia or neurological or psychiatric pathology.
* Patients with a transient global amnesia according to the criteria of Hodges and Warlow (1990) in the acute phase (i.e. within 24 hours after the onset of the stroke), accompanied by a trusted person
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in another study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding
* Presence of a focal neurological pathology that may explain the symptoms, history of epilepsy or psychiatric disorders.
* Hypersensitivity to iodinated contrast media.
* Known allergy to 18-FDG.

Non-inclusion criteria concerning control subjects:

* Presence of disorders on neurological assessment
* Presence of cognitive disorders on the neuropsychological assessment (z-score <-1.65 on the RBANS or on the Stroop test).

Exclusion criteria for the target population:

• Patients will be excluded after the 1st neuropsychological assessment if episodic memory tests show complete recovery from anterograde amnesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with a transient global amnesia according to the criteria of Hodges and Warlow (1990) in the acute phase (i.e. within 24 hours after the onset of the stroke), accompanied by a trusted person and admitted to the SAU of the CHU de Nîmes, plus a group of healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Storage and retrieval capacities of information with a strong emotional valence in patients compared to healthy controls | Day 0
  International Affective Picture System (IAPS): number of correctly memorized images of each type of emotional content (15 positive, 15 negative and 15 neutral).
Ability to judge the degree of activation and emotional value associated with images | Day 0
  Self Assessment Manikin (SAM)

SECONDARY OUTCOMES:
Change in storage and retrieval capacities of information with a strong emotional valence in patients from baseline | Day 3
  International Affective Picture System (IAPS): number of correctly memorized images of each type of emotional content (15 positive, 15 negative and 15 neutral).
Change in storage and retrieval capacities of information with a strong emotional valence in patients from baseline | Month 3
  International Affective Picture System (IAPS): number of correctly memorized images of each type of emotional content (15 positive, 15 negative and 15 neutral).
Classification of event triggering transient global amnesia | Day 0
  Psychological/physiological
Anxiety | Day 0
  Hamilton Scale: where score = 7 is absence of depression; 8-15 is minor depression and 16 or more is severe depression
Depression | Day 0
  Beck Depression Scale
Mood | Day 0
  Befindlichkeits Skala Mood Scale
C-score of the Groupe de REflexion pour l'Evaluation des Fonctions Exécutives (GREFEX) version of Stroop Test between patients and healthy control | Day 0
  Stroop Test
Repeatable Battery for the Assessment of Neuropsychological Status between patients and healthy control | Day 0
  Repeatable Battery for the Assessment of Neuropsychological Status: 10 subtests combined into 5 index scores and 1 total score.
Identification of hypometablic zones by PET compared to age- and sex-matched controls | Day 0
  Visual analysis of hippocampus and other topographies (Z-score); Statistical Parametric Mapping 12

CONTACTS AND LOCATIONS:
Overall Officials: Eric THOUVENOT, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France